CLINICAL TRIAL: NCT03888716
Title: A Phase Ia/Ib, Multiple-site Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of KL1333 After a Single and Multiple Ascending Oral Doses in Healthy Subjects and Patients With Primary Mitochondrial Disease
Brief Title: A Phase Ia/Ib, SAD and MAD Study of of KL1333 in Healthy Subjects and Patients With Primary Mitochondrial Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abliva AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KL1333 2018-102
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Mitochondrial Diseases; Mitochondrial Respiratory Chain Deficiencies; MELAS Syndrome; Mitochondrial Myopathies
Keywords: Mitochondrial Diseases; Mitochondrial Respiratory Chain Deficiencies; MELAS Syndrome; Mitochondrial Myopathies; Kearns-Sayre Syndrome; Ophthalmoplegia, Chronic Progressive External
MeSH Terms: conditions — Mitochondrial Diseases; MELAS Syndrome; Mitochondrial Myopathies; Kearns-Sayre Syndrome; Ophthalmoplegia, Chronic Progressive External

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KL1333 (Experimental): 25 and 100 mg KL1333 encapsulated tablets for daily oral dosing
  Interventions: Drug: KL1333
- Matching placebo (Placebo Comparator): 25 and 100 mg KL placebo encapsulated tablets for daily oral dosing
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: KL1333 — 25 and 100 mg KL1333 encapsulated tablets
  Arms: KL1333
Drug: Placebo Oral Tablet — 25 and 100 mg placebo encapsulated tablets
  Arms: Matching placebo

SUMMARY:
This will be a double blind, randomised, placebo controlled, single and multiple oral dose study conducted in 3 parts: Part A, Part B and Part C. Part A and Part B include healthy volunteers only and will be completed before Part C including patients with primary mitochondrial disease will be initiated. The starting dose in the first cohort of Part A will be 25 mg. The dose level in the additional cohorts will be decided following review of data of the previous cohorts.

DETAILED DESCRIPTION:
Part A: Eight healthy subjects will be studied in a single cohort (Group A1). Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will participate in 2 treatment periods, fasting or after consuming a standard high-fat breakfast. For each treatment period, subjects will reside at the Phase I clinical site from Days 1 to 3 (48 hours postdose). Subjects will return to the clinical site for outpatient visits on Days 4 and 5. There will be at least a 10 day washout between doses Additional single-dose cohorts may be enrolled based on data obtained from either Parts A or B.

Part B: Sixteen healthy subjects will be studied in 2 cohorts (Groups B1 and B2), with each cohort consisting of 8 subjects. Following review of safety, tolerability, and PK data, up to 3 additional dose cohorts of healthy subjects may be added to further explore the PK, safety, and tolerability of KL1333. Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. All subjects will participate in 1 treatment period and will reside at the Phase I clinical site from Days -1 to 12 (48 hours post final dose). Subjects will return to the clinical site for outpatient visits on Days 13 and 14. On Day 1, 6 subjects will be randomised to receive KL1333 and 2 subjects will be randomised to receive placebo. Subjects will return for a Follow-up visit on Day 15, 5 days after their final dose.

Part C: A total of 8 patients diagnosed with any mitochondrial disease will be enrolled in this part of the study. Part C may start after the dose selection conference has been completed for the final cohort of Part B, at a daily dose no higher than the highest well-tolerated dose in Part B. Potential study patients will be screened to assess their eligibility to enter the study within 35 days prior to the first dose administration. Patients will reside at the clinical site from Days -1 to 2 and Days 10 to 11 and return to the clinical site for outpatient visits on Days 4 and 8. It is planned for patients to receive study drug once daily on Days 1 to 10. Patients will return for a Follow-up visit on Day 15, 5 days after their final dose.

ELIGIBILITY:
Inclusion Criteria (selected):

Healthy subjects and patients with mitochondrial disease must satisfy all of the following criteria at the Screening visit unless otherwise stated:

1. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
2. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
3. Able to perform all protocol-specified assessments and comply with the study visit schedule.

   Additional inclusion criteria for healthy subjects:
4. Males or females, of any race, between 18 and 65 years of age, inclusive.
5. Weight ≥50 kg and body mass index between 18.0 and 32.0 kg/m2, inclusive.
6. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhaemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening and Check in as assessed by the Investigator.

   Additional inclusion criteria for patients with mitochondrial disease:
7. Males or females, of any race, between 18 and 75 years of age, inclusive.
8. Body mass index between 15.0 and 32.0 kg/m2, inclusive.
9. Any mitochondrial disease that has been genetically confirmed.
10. Clinically stable, apart from symptoms associated with the diagnosis of mitochondrial disease, as determined by medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations at Screening and Check-in as assessed by the Investigator.

Exclusion Criteria (selected):

Healthy subjects and patients with mitochondrial disease will be excluded from the study if they satisfy any of the following criteria at the Screening visit unless otherwise stated:

1. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, including KL1333 or its excipients, unless approved by the Investigator.
2. History of gastroesophageal reflux disease, gastric erosions, peptic ulcer disease, or gastrointestinal bleeding episodes.
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs including cholecystectomy (uncomplicated appendectomy and hernia repair will be allowed).
4. History of malignancy of any organ system other than localised basal cell carcinoma of the skin, treated or untreated, within 5 years prior to Screening, regardless of whether there is evidence of local recurrence or metastases.
5. History of clinically significant illness (except for mitochondrial disease in the patients in Part C) or surgery within 4 weeks prior to Screening, as determined by the Investigator.
6. History of alcoholism or drug/chemical abuse within 2 years prior to Screening.
7. Alcohol consumption of >28 units per week for males and >21 units per week for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
8. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check in.
9. Positive hepatitis panel and/or positive human immunodeficiency virus test

Additional exclusion criteria for patients with mitochondrial disease:

1. Use of idebenone or medications (prescription or nonprescription) that have effects on metabolism or unknown binding sites (eg, vitamin E, co-enzyme 10, arginine) within 35 days or 5 half-lives, whichever is longer, prior to the first dose.
2. Use of prescription drugs within 14 days prior to dosing, with the exception of established therapy for mitochondrial disease and the treatment of associated disorders that has been stable for at least 7 days prior to the first dose, as approved by the Medical Monitor and Investigator, in consultation with the Sponsor.
3. Uncontrolled diabetes mellitus, as determined by the Investigator. Creatinine clearance <45 mL/min as calculated by the Cockcroft-Gault equation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Safety: incidence and severity of AEs | Day 15
Safety: incidence of laboratory abnormalities, based on haematology, clinical chemistry, and urinalysis test results | Day 15
Safety: 12 lead ECG parameters | Day 15
Safety: Number of participants with clinically significant abnormal vital signs measurements | Day 15
Safety: Number of participants with clinically significant abnormal physical examinations | Day 15

SECONDARY OUTCOMES:
PK: area under the curve, AUC0 ∞ | Day 1
PK: AUC over a dosing interval (AUC0 τ) | Days 1 and 10
PK: temporal change parameter (TCP; AUC0 τ/AUC0-∞) | Days 1 and 10
PK: Cmax | Day 1
PK: time of the Cmax (Tmax) | Day 1
PK: minimum observed plasma concentration (Cmin) | Days 1 and 10
PK: apparent plasma terminal elimination half life (t1/2) | Days 1 and 10
PK: mean residence time (MRT) | Days 1 and 10
PK: apparent total plasma clearance (CL/F) | Days 1 and 10
PK: apparent volume of distribution during the terminal phase (Vz/F) | Days 1 and 10

OTHER OUTCOMES:
NAD+/NADH concentrations and ratio (part B and C) | Days 10 and 15
  Biomarker
FGF21 and GDF15 concentrations (part B and C) | Days 10 and 15
  Biomarker
Lactate/pyruvate concentrations and ratio (part B and C) | Days 10 and 15
  Biomarker
Newcastle Mitochondrial Disease Adult Scale (NMDAS) (part C) | Day 10
  Assessment of mitochondrial disease. The NMDAS is a validated clinical rating scale designed to capture the natural history of mitochondrial disease. The NMDAS includes 3 domains: current function, system specific involvement, and current clinical, assessed on 6-point Likert-type scale from 0 to 5, as well as a fourth section including a score for the 12-Item Short Form Survey-Version 2.
Clinician Global Impression (CGI) (part C) | Day 10
  Assessment of illness severity, global improvement or change, and therapeutic response.The CGI is a 3-item observer-rated scale that measures illness severity, global improvement or change, and therapeutic response. The CGI is rated on a 7-point Likert-type scale, with the severity of illness scale using a range of responses from 1 (normal) to 7 (amongst the most severely ill patients).
Patient Global Impression-Improvement (PGI-I) (part C) | Day 10
  Patient reported assessment of severity of illness. The PGI-I is a patient-rated scale using a 7-point Likert-type scale, with the severity of illness scale using a range of responses from 1 (normal) to 7 (amongst the most severely ill patients). An item about the patient's worst symptom will be included in the assessment for this study.
Daily Fatigue Impact Severity (D-FIS) (part C) | Day 10
  Assessment of fatigue. The D-FIS is a patient-rated scale developed to assess the symptom of fatigue as part of an underlying chronic disease or condition. The D-FIS includes 8 items assessed on 5-point Likert-type scale from 0 (no problem) to 4 (extreme problem).
Quality of Life in Neurological Disorders Fatigue Scale (Neuro-QoL Fatigue) (part C) | Day 10
  Assessment of fatigue. The Neuro-QoL Fatigue is one of several scales that make up the Quality of Life in Neurological Disorders measurement system. It is a reliable and validated brief 19-item survey of fatigue, completed by the subject, with a recall period of the past 7 days. The 19 items are scored from 1 (never) to 5 (always) and consequently, Neuro-QoL Fatigue total scores range from 19 to 95, with higher scores indicating greater fatigue and greater impact of mitochondrial disease on activities.
30 Second Sit-to-Stand Test (part C) | Day 10
  Test

CONTACTS AND LOCATIONS:
Overall Officials: Matilda Hugerth, MSc, Study Director — Abliva AB
Locations (2):
- United Kingdom (2):
  - Covance Leeds, Leeds, West Yorkshire
  - UCL, London

IPD SHARING:
Plan to Share IPD: No
According to EMA rules.